CLINICAL TRIAL: NCT01590654
Title: A Double-Blind, Randomized, Placebo-Controlled, Single and Multiple-Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antiviral Activity of GS-9620 in Virologically Suppressed Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Study Evaluating GS-9620 in Virologically Suppressed Subjects With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-283-0102
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis B
Keywords: Hepatitis; Hepatitis B; Hepatitis B Virus; HBV; GS-9620; Toll-like receptor (TLR)-7 Agonist
MeSH Terms: conditions — Hepatitis B; Hepatitis | interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 0.3mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 1mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 2mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 4mg GS-9620 (Experimental)
  Interventions: Drug: Single Ascending Dose (SAD) Cohorts GS-9620
- 0.3mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts GS-9620
- 1mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts GS-9620
- 2mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts GS-9620
- 4mg GS-9620 QW x 2 doses (Experimental)
  Interventions: Drug: Multiple Ascending Dose (MAD) Cohorts GS-9620

INTERVENTIONS:
Drug: Single Ascending Dose (SAD) Cohorts GS-9620 — This study will enroll cohorts of 6 eligible, unique subjects per cohort, randomized to either active drug or placebo (5:1) within each cohort. Subjects in Single Ascending Dose (SAD) Cohorts will receive a single dose of GS-9620.
  Arms: 0.3mg GS-9620; 1mg GS-9620; 2mg GS-9620; 4mg GS-9620
Drug: Multiple Ascending Dose (MAD) Cohorts GS-9620 — This study will enroll cohorts of 6 eligible, unique subjects per cohort, randomized to either active drug or placebo (5:1) within each cohort. Subjects in Multiple Ascending Dose (MAD) Cohorts will receive GS-9620 once weekly for two weeks (QW x 2 doses).
  Arms: 0.3mg GS-9620 QW x 2 doses; 1mg GS-9620 QW x 2 doses; 2mg GS-9620 QW x 2 doses; 4mg GS-9620 QW x 2 doses

SUMMARY:
Dose cohorts may be dosed with one of up to 4 possible total weekly doses (0.3 mg, 1 mg, 2 mg, 4 mg). Dose escalation or repetition will be governed by pre-specified safety and activity rules. Subjects will be confined on days 1-3 and/or days 8-10. Follow-up visits are required periodically through day 43. Subjects with sustained reductions in HbsAg will be requested to return for additional follow-up follow-up visits at 3 and 6 months post last dose. Study procedures involve blood draws for pharmacokinetic, pharmacodynamic, virologic, and safety assessments

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection for ≥ 6 months
* Currently on treatment with at least 1 HBV approved oral drug (i.e. lamivudine, telbivudine, entecavir, adefovir, tenofovir) ≥ 3 months prior to screening
* HBsAg ≥ 250 IU/mL
* HBV DNA at below the level of quantitation (BLQ; to be confirmed at screening)
* Absence of extensive bridging fibrosis (Metavir 3 or greater)or cirrhosis
* Creatinine clearance ≥ 70 mL/min

Exclusion Criteria:

* Co-infection with hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV
* History of Gilberts disease
* Laboratory parameters not within defined thresholds for leukopenia, neutropenia, anemia, thrombocytopenia, thyroid-stimulating hormone (TSH), or other evidence of hepatic decompensation
* Diagnosis of autoimmune disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), malignancy, hemoglobinopathy, retinal disease, or patients who are immunosuppressed
* Evidence of hepatocellular carcinoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events in single and multiple oral doses of GS-9620 | Periodically Day 1 to 6 months
  Assessments include adverse events, laboratory abnormalities, 12-lead ECG abnormalities and interval measurements, and vital signs measurements

SECONDARY OUTCOMES:
Assessment of plasma drug concentrations of GS-9620 using non-compartmental methods | Day 1 and Day 8
  SAD and MAD Cohorts:serial blood samples will be collected on Day 1 at 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, and 96 hours post-dose.
  Mad Cohorts: serial blood samples will also be collected on Day 8 at 0 (pre-dose), , 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, and 24 hours post-dose.
Measurement of pharmacodynamic markers (cytokines and interferon-stimulated genes [ISGs]) | Days 1, 2, 3, 5, 8
  Single ascending dose (SAD) Cohorts: Whole blood and serum for pharmacodynamic (PD) assessments (RNA and cytokine analysis) will be drawn on Day 1 at pre-dose, 8, 24 and 48 hours post-dose, and on Days 5 and Day 8
  Multiple ascending dose (MAD) Cohorts: Whole blood and serum for PD assessments (RNA and cytokine analysis) will be drawn on Day 1: Pre-dose and 8 hours Postdose, Day 2, Day 3, and Day 5 Day 8: Pre-dose and 8 hours Post-dose, Day 9, 10, 12, and Day 15
Reduction of hepatitis B (HBV) viral load from baseline | Screening, Baseline, Day 8 or 15
  SAD cohort: HBsAg+ levels will be drawn at Day 1: Pre-dose, Day 2, 3, 5, 8 and both Follow-up Visits.
  MAD cohorts: HBsAg+ levels will be drawn at Day 1: Pre-dose, Day 2, 3, 5, Day 8: Pre-Dose, 9, 10, 15, and both Follow-Up Visits.

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Massetto, M.D., Study Director — Gilead Sciences
Locations (20):
- United States (9):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Indiana University Medical Center, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Weill Cornell Medical College, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (5):
  - Nepean Hospital, Department of ID, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Monash University, Dept. of Medicine, Clayton, Victoria
  - Alfred Hospital, Department of Gastroenterology, Melbourne, Victoria
  - Royal Perth Hospital, Nedlands, Western Australia
- Canada (3):
  - University of Calgary, Heritage Medical Research Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Algorithme Pharma, Inc., Laval, Quebec
- Aukland Clinical Studies, Grafton, Aukland, New Zealand
- South Korea (2):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul